CLINICAL TRIAL: NCT04625725
Title: A Phase III Randomized, Double-blind, Placebo-controlled, Multi-center Study in Adults to Determine the Safety and Efficacy of AZD7442, a Combination Product of Two Monoclonal Antibodies (AZD8895 and AZD1061), for Pre-exposure Prophylaxis of COVID-19.
Brief Title: Phase III Double-blind, Placebo-controlled Study of AZD7442 for Pre-exposure Prophylaxis of COVID-19 in Adult.
Acronym: PROVENT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: D8850C00002; 2020-004356-16 (EudraCT Number)
Record Dates: First submitted 2020-11-10; First posted 2020-11-12 (Actual); Results first posted 2022-12-20 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: COVID-19
Keywords: Pre-exposure Prophylaxis of COVID-19
MeSH Terms: conditions — COVID-19 | interventions — cilgavimab and tixagevimab drug combination; cilgavimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- AZD7442 (Experimental): Approximately 5150 participants will be randomized in a 2:1 ratio
  • Arm 1 (n=approximately 3433) will receive a single dose (× 2IM injections) of 300 mg of AZD7442
  Interventions: Drug: AZD7442
- Placebo (Placebo Comparator): Approximately 5150 participants will be randomized in a 2:1 ratio
  • Arm 2 (n=approximately 1717) will receive saline placebo
  Interventions: Drug: Placebo
- Sub-study AZD7442 Arm 1 (Experimental): Approximately 500 participants will receive AZD7442 in the repeat dose sub-study.
  -Sub-study Arm 1 (~ 12 month repeat dose interval): Participants who received AZD7442 300 mg IM on Day 1 of the parent study will receive a second dose of AZD7442 300mg IM on sub-study Day 1.
  Interventions: Drug: AZD7442
- Sub-study AZD7442 Arm 2 (Experimental): Approximately 500 participants will receive AZD7442 in the repeat dose sub-study.
  -Sub-study Arm 2(~ 6 month repeat dose interval): Participants who received placebo on Day 1 of the parent study will receive their first dose of AZD7442 300mg IM on sub-study Day1 followed by a second dose on sub-study Day 183.
  Interventions: Drug: AZD7442
- Sub-study AZD7442 Arm 3 (Experimental): A subset of Arm 1 and Arm 2 participants who will receive additional doses of AZD7442, 600mg, at Day 183 and Day 366 of the sub-study.
  Interventions: Drug: AZD7442

INTERVENTIONS:
Drug: AZD7442 — * Single dose (× 2IM injections) of 300 mg of AZD7442 on parent study Day 1.
  * Single dose (× 2IM injections) of 300 mg of AZD7442 on sub-study Day 1.
  * Single dose (× 2IM injections) of 300 mg of AZD7442 on sub-study Day 183.
  * Single dose (x 2IM injections) of 600mg of AZD7442 on sub-study Day 183 and Day 366
  Other Names: Combination of 2mAbs(AZD8895 and AZD1061)
  Arms: AZD7442; Sub-study AZD7442 Arm 1; Sub-study AZD7442 Arm 2; Sub-study AZD7442 Arm 3
Drug: Placebo — Single dose (× 2IM injections) of saline placebo on parent study Day 1.
  Arms: Placebo

SUMMARY:
This study will assess the safety and efficacy of a single dose of AZD7442(× 2 IM injections) compared to placebo for the prevention of COVID-19.

DETAILED DESCRIPTION:
SARS-CoV-2 is the causative agent of the ongoing COVID-19 pandemic that, as of 29 September 2020, has resulted in a high death toll to date. Unlike the majority of coronaviruses that cause mild disease in humans and animals, SARS-CoV-2 can replicate in the lower respiratory tract to cause acute respiratory distress syndrome and fatal pneumonia. Effective interventions to prevent or treat COVID-19 remain limited in number and clinical experience is limited. Clinical management is limited to supportive care, consequently overwhelming resources of healthcare systems around the world. As a response to the ongoing pandemic, AstraZeneca is developing mAbs to the SARS-CoV-2 S protein. The SARS-CoV-2 spike protein contains the virus's RBD, which enables the virus to bind to receptors on human cells. By targeting this region of the virus's spike protein, antibodies can block the virus's attachment to human cells, and, therefore, is expected to block infection. Amino acid substitutions have been introduced into the antibodies to both extend their half-lives, which should prolong their potential prophylactic benefit, and decrease Fc effector function in order to decrease the potential risk of antibody-dependent enhancement of disease. AZD7442, a combination of 2 of these mAbs (AZD8895 and AZD1061), is being evaluated for administration to prevent and/or treat COVID-19. There is currently one completed and 2 ongoing Phase I studies with AZD7442.

-The Provent repeat dose open-label sub-study is initiated to assess the safety, PK and immunogenicity of repeat doses of AZD7442 in participants currently enrolled in the Provent study who may benefit from repeat dose of AZD7442.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age at the time of signing the informed consent
2. Can benefit from passive immunization with antibodies
3. Medically stable
4. Negative result from point of care SARS-CoV-2 serology testing at screening
5. Contraceptive used by women of child bearing potential, condom used by men
6. Able to understand and comply with study requirements/procedures based on the assessment of the investigator

Sub-study Inclusion criteria which are additional to those in parent study are as follows:

* The participant has been randomized, dosed, and is ongoing in the PROVENT parent study and is 12±2 months post first dose of blinded IMP.
* If one or more of the following apply:

  1. Immunocompromised and/or may be at increased risk for an inadequate immune response to a COVID-19 vaccine.
  2. In the opinion of the Investigator, are at increased risk and would benefit from a repeat dose of AZD7442.
* Documented negative SARS-CoV-2 RT-PCR test collected ≤ 3 days prior to sub-study Day 1 or a negative rapid SARS-CoV-2 antigen test at screening.

Exclusion Criteria:

1. Significant infection or other acute illness, including fever >100°F (>37.8°C) on the day prior to or day of randomization.
2. History of laboratory-confirmed SARS-CoV-2 infection or any positive SARS-CoV-2 result based on available data at screening.
3. History of infection with severe acute respiratory syndrome (SARS) or Middle East respiratory syndrome (MERS).
4. Known history of allergy or reaction to any component of the study drug formulation.
5. Previous hypersensitivity, infusion-related reaction, or severe adverse reaction following administration of a mAb.
6. Any prior receipt of investigational or licensed vaccine or other mAb/biologic indicated for the prevention of SARS-CoV-2 or COVID-19 or expected receipt during the period of study follow-up.
7. Bleeding disorder or prior history of significant bleeding or bruising following IM injections or venepuncture.
8. Any other significant disease, disorder, or finding. that may significantly increase the risk to the participant because of participation in the study, affect the ability of the participant to participate in the study, or impair interpretation of the study data.
9. Receipt of any IMP in the preceding 90 days or expected receipt of IMP during the period of study follow-up, or concurrent participation in another interventional study
10. Currently pregnant or breastfeeding.
11. Blood drawn in excess of a total of 450 mL (1 unit) for any reason within 30 days prior to randomization.
12. Employees of the Sponsor involved in planning, executing, supervising, or reviewing the AZD7442 program,, clinical study site staff, or any other individuals involved with the conduct of the study, or immediate family members of such individuals.
13. In nations, states, or other jurisdictions that for legal or ethical reasons bar the enrollment of participants who lack capacity to provide their own informed consent, such subjects are excluded.

Sub-study Exclusion criteria are as follows:

1. Patient have received a COVID-19 vaccination ≤ 14 days before sub-study Day1 or plan to receive a COVID-19 vaccination ≤ 14 days after sub-study Day1. (Such participants can subsequently be included in the study once they have reached >14 days after their last dose of vaccine).
2. Patient have two or more untreated cardiac risk factors or suspected unstable cardiac disease.
3. Judgment by the Investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions, and requirements.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5197 (Actual)
Dates: Start 2020-11-21 (Actual); Primary Completion 2022-08-16 (Actual); Study Completion 2023-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Myron Levin, MD, Principal Investigator — AstraZeneca
Locations (83):
- United States (56):
  - Research Site, Birmingham, Alabama
  - Research Site, Tempe, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Cerritos, California
  - Research Site, Fresno, California
  - Research Site, Garden Grove, California
  - Research Site, Huntington Beach, California
  - Research Site, Lancaster, California
  - Research Site, Modesto, California
  - Research Site, Victorville, California
  - Research Site, Westminster, California
  - Research Site, Hartford, Connecticut
  - Research Site, Middlebury, Connecticut
  - Research Site, Clearwater, Florida
  - Research Site, Coral Springs, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Lauderdale Lakes, Florida
  - Research Site, Miami, Florida
  - Research Site, Ormond Beach, Florida
  - Research Site, Pompano Beach, Florida
  - Research Site, Wesley Chapel, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Columbus, Georgia
  - Research Site, Conyers, Georgia
  - Research Site, Marietta, Georgia
  - Research Site, Honolulu, Hawaii
  - Research Site, Chicago, Illinois
  - Research Site, Hazel Crest, Illinois
  - Research Site, Quincy, Illinois
  - Research Site, Evansville, Indiana
  - Research Site, Noblesville, Indiana
  - Research Site, Wichita, Kansas
  - Research Site, Minneapolis, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Omaha, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Albuquerque, New Mexico
  - Research Site, Jamaica, New York
  - Research Site, Ridgewood, New York
  - Research Site, The Bronx, New York
  - Research Site, Greensboro, North Carolina
  - Research Site, Columbus, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Summerville, South Carolina
  - Research Site, Rapid City, South Dakota
  - Research Site, Austin, Texas
  - Research Site, El Paso, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Shenandoah, Texas
  - Research Site, Sugar Land, Texas
  - Research Site, Layton, Utah
  - Research Site, Alexandria, Virginia
  - Research Site, Chesapeake, Virginia
  - Research Site, Tacoma, Washington
- Belgium (5):
  - Research Site, Alken
  - Research Site, Brussels
  - Research Site, Gozée
  - Research Site, Namur
  - Research Site, Wetteren
- France (9):
  - Research Site, Clermont-Ferrand
  - Research Site, Dijon
  - Research Site, La Roche S/ Yon Cedex 9
  - Research Site, Lille
  - Research Site, Limoges
  - Research Site, Nantes
  - Research Site, Paris
  - Research Site, Saint-Etienne
  - Research Site, Tours
- Spain (4):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Marbella (Málaga)
  - Research Site, Pozuelo de Alarcón
- United Kingdom (9):
  - Research Site, Bournemouth
  - Research Site, Enfield
  - Research Site, Hayle
  - Research Site, London
  - Research Site, Preston
  - Research Site, Rochdale
  - Research Site, Salford
  - Research Site, Torpoint
  - Research Site, Wakefield

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Background] Antonia SJ, Villegas A, Daniel D, Vicente D, Murakami S, Hui R, Kurata T, Chiappori A, Lee KH, de Wit M, Cho BC, Bourhaba M, Quantin X, Tokito T, Mekhail T, Planchard D, Kim YC, Karapetis CS, Hiret S, Ostoros G, Kubota K, Gray JE, Paz-Ares L, de Castro Carpeno J, Faivre-Finn C, Reck M, Vansteenkiste J, Spigel DR, Wadsworth C, Melillo G, Taboada M, Dennis PA, Ozguroglu M; PACIFIC Investigators. Overall Survival with Durvalumab after Chemoradiotherapy in Stage III NSCLC. N Engl J Med. 2018 Dec 13;379(24):2342-2350. doi: 10.1056/NEJMoa1809697. Epub 2018 Sep 25. PMID 30280658
- [Background] CDC. (Centers for Disease Control and Prevention). Coronavirus Disease 2019 (COVID-19), Symptoms of Coronavrus. https://www.cdc.gov/coronavirus/2019-ncov/symptomstesting/symptoms.html. Published 2020. Accessed 01 July 2020.
- [Background] Domachowske JB, Khan AA, Esser MT, Jensen K, Takas T, Villafana T, Dubovsky F, Griffin MP. Safety, Tolerability and Pharmacokinetics of MEDI8897, an Extended Half-life Single-dose Respiratory Syncytial Virus Prefusion F-targeting Monoclonal Antibody Administered as a Single Dose to Healthy Preterm Infants. Pediatr Infect Dis J. 2018 Sep;37(9):886-892. doi: 10.1097/INF.0000000000001916. PMID 29373476
- [Background] Furer V, Rondaan C, Heijstek MW, Agmon-Levin N, van Assen S, Bijl M, Breedveld FC, D'Amelio R, Dougados M, Kapetanovic MC, van Laar JM, de Thurah A, Landewe RB, Molto A, Muller-Ladner U, Schreiber K, Smolar L, Walker J, Warnatz K, Wulffraat NM, Elkayam O. 2019 update of EULAR recommendations for vaccination in adult patients with autoimmune inflammatory rheumatic diseases. Ann Rheum Dis. 2020 Jan;79(1):39-52. doi: 10.1136/annrheumdis-2019-215882. Epub 2019 Aug 14. PMID 31413005
- [Background] Coronaviridae Study Group of the International Committee on Taxonomy of Viruses. The species Severe acute respiratory syndrome-related coronavirus: classifying 2019-nCoV and naming it SARS-CoV-2. Nat Microbiol. 2020 Apr;5(4):536-544. doi: 10.1038/s41564-020-0695-z. Epub 2020 Mar 2. PMID 32123347
- [Background] Griffin MP, Khan AA, Esser MT, Jensen K, Takas T, Kankam MK, Villafana T, Dubovsky F. Safety, Tolerability, and Pharmacokinetics of MEDI8897, the Respiratory Syncytial Virus Prefusion F-Targeting Monoclonal Antibody with an Extended Half-Life, in Healthy Adults. Antimicrob Agents Chemother. 2017 Feb 23;61(3):e01714-16. doi: 10.1128/AAC.01714-16. Print 2017 Mar. PMID 27956428
- [Background] Griffin MP, Yuan Y, Takas T, Domachowske JB, Madhi SA, Manzoni P, Simoes EAF, Esser MT, Khan AA, Dubovsky F, Villafana T, DeVincenzo JP; Nirsevimab Study Group. Single-Dose Nirsevimab for Prevention of RSV in Preterm Infants. N Engl J Med. 2020 Jul 30;383(5):415-425. doi: 10.1056/NEJMoa1913556. PMID 32726528
- [Background] Lamb EJ, Levey AS, Stevens PE. The Kidney Disease Improving Global Outcomes (KDIGO) guideline update for chronic kidney disease: evolution not revolution. Clin Chem. 2013 Mar;59(3):462-5. doi: 10.1373/clinchem.2012.184259. No abstract available. PMID 23449698
- [Background] Li F. Structure, Function, and Evolution of Coronavirus Spike Proteins. Annu Rev Virol. 2016 Sep 29;3(1):237-261. doi: 10.1146/annurev-virology-110615-042301. Epub 2016 Aug 25. PMID 27578435
- [Background] Morand EF, Furie RA. Anifrolumab in Systemic Lupus Erythematosus. Reply. N Engl J Med. 2020 Apr 23;382(17):1666. doi: 10.1056/NEJMc2002191. No abstract available. PMID 32320577
- [Background] Poland GA, Ovsyannikova IG, Kennedy RB. Personalized vaccinology: A review. Vaccine. 2018 Aug 28;36(36):5350-5357. doi: 10.1016/j.vaccine.2017.07.062. Epub 2017 Jul 31. PMID 28774561
- [Background] Robbie GJ, Criste R, Dall'acqua WF, Jensen K, Patel NK, Losonsky GA, Griffin MP. A novel investigational Fc-modified humanized monoclonal antibody, motavizumab-YTE, has an extended half-life in healthy adults. Antimicrob Agents Chemother. 2013 Dec;57(12):6147-53. doi: 10.1128/AAC.01285-13. Epub 2013 Sep 30. PMID 24080653
- [Background] Wagner A, Weinberger B. Vaccines to Prevent Infectious Diseases in the Older Population: Immunological Challenges and Future Perspectives. Front Immunol. 2020 Apr 23;11:717. doi: 10.3389/fimmu.2020.00717. eCollection 2020. PMID 32391017
- [Background] WHO. WHO Coronavirus Disease (COVID-19) Dashboard. 2020a.
- [Background] WHO. WHO R&D Blueprint COVID-19 Therapeutic Trial Synopsis Draft 18 February 2020. https://www.who.int/blueprint/priority-diseases/key-action/COVID19_Treatment_Trial_Design_Master_Protocol_synopsis_Final_18022020.pdf. Published 2020b. Accessed 25 September 2020.
- [Background] Zhou P, Yang XL, Wang XG, Hu B, Zhang L, Zhang W, Si HR, Zhu Y, Li B, Huang CL, Chen HD, Chen J, Luo Y, Guo H, Jiang RD, Liu MQ, Chen Y, Shen XR, Wang X, Zheng XS, Zhao K, Chen QJ, Deng F, Liu LL, Yan B, Zhan FX, Wang YY, Xiao GF, Shi ZL. A pneumonia outbreak associated with a new coronavirus of probable bat origin. Nature. 2020 Mar;579(7798):270-273. doi: 10.1038/s41586-020-2012-7. Epub 2020 Feb 3. PMID 32015507
- [Background] Zimmermann P, Curtis N. Factors That Influence the Immune Response to Vaccination. Clin Microbiol Rev. 2019 Mar 13;32(2):e00084-18. doi: 10.1128/CMR.00084-18. Print 2019 Mar 20. PMID 30867162
- [Background] Zou G. A modified poisson regression approach to prospective studies with binary data. Am J Epidemiol. 2004 Apr 1;159(7):702-6. doi: 10.1093/aje/kwh090. PMID 15033648
- [Derived] Ustianowski A, Levin MJ, De Wit S, Launay O, Veekmans B, Rampling T, Sullivan JG, Vishnepolsky M, Wijewardane P, Fawadleh Y, Zhang H, Li M, Wickramarachchi D, Sharbaugh A, Beavon R, Thissen J, Hirao L, Dzutseva V, Seegobin S, Streicher K, Kiazand A, Esser MT, Chang LJ, Perez JL, Cohen TS. Safety and Pharmacokinetics of Repeat Dosing of Long-Acting SARS-CoV-2 Antibodies Tixagevimab/Cilgavimab (AZD7442): Results from the PROVENT Sub-study. Clin Drug Investig. 2026 Jan 16. doi: 10.1007/s40261-025-01515-x. Online ahead of print. PMID 41545648
- [Derived] Levin MJ, Ustianowski A, De Wit S, Beavon R, Thissen J, Seegobin S, Dey K, Near KA, Streicher K, Kiazand A, Esser MT. Efficacy, Safety, and Pharmacokinetics of AZD7442 (Tixagevimab/Cilgavimab) for Prevention of Symptomatic COVID-19: 15-Month Final Analysis of the PROVENT and STORM CHASER Trials. Infect Dis Ther. 2024 Jun;13(6):1253-1268. doi: 10.1007/s40121-024-00970-x. Epub 2024 May 4. PMID 38703336
- [Derived] Tuffy KM, Ahani B, Aksyuk AA, Avila M, Brady T, Kijak GH, Koh G, Levin MJ, Roe TL, Schuko N, Thissen J, Ustianowski A, Zhang T, Kelly EJ, Streicher K. Breakthrough SARS-CoV-2 Infections in the PROVENT Prevention Trial Were Not Associated With AZD7442 (Tixagevimab/Cilgavimab) Resistant Variants. J Infect Dis. 2023 Oct 18;228(8):1055-1059. doi: 10.1093/infdis/jiad210. PMID 37280116
- [Derived] Hirsch C, Park YS, Piechotta V, Chai KL, Estcourt LJ, Monsef I, Salomon S, Wood EM, So-Osman C, McQuilten Z, Spinner CD, Malin JJ, Stegemann M, Skoetz N, Kreuzberger N. SARS-CoV-2-neutralising monoclonal antibodies to prevent COVID-19. Cochrane Database Syst Rev. 2022 Jun 17;6(6):CD014945. doi: 10.1002/14651858.CD014945.pub2. PMID 35713300
- [Derived] Levin MJ, Ustianowski A, De Wit S, Launay O, Avila M, Templeton A, Yuan Y, Seegobin S, Ellery A, Levinson DJ, Ambery P, Arends RH, Beavon R, Dey K, Garbes P, Kelly EJ, Koh GCKW, Near KA, Padilla KW, Psachoulia K, Sharbaugh A, Streicher K, Pangalos MN, Esser MT; PROVENT Study Group. Intramuscular AZD7442 (Tixagevimab-Cilgavimab) for Prevention of Covid-19. N Engl J Med. 2022 Jun 9;386(23):2188-2200. doi: 10.1056/NEJMoa2116620. Epub 2022 Apr 20. PMID 35443106
- See also: CSP redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8850C00002&attachmentIdentifier=15030b78-ad9f-4ab2-9cca-b0e90eda0fda&fileName=CSP_redacted.pdf&versionIdentifier=
- See also: SAP redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8850C00002&attachmentIdentifier=c5bf455f-561e-44e0-9b5d-fc359b919e81&fileName=SAP_redacted.pdf&versionIdentifier=
- See also: CSR synopsis redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8850C00002&attachmentIdentifier=7fef0350-165b-4990-b0dd-746411144169&fileName=CSR_synopsis_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- AZD7442: 300 mg (AZD8895 and AZD1061)
- Placebo: Saline Placebo
- Group1: 2 doses of AZD7442 300mg, 10-14 months schedule
- Group 2: 2 doses ofAZD7442 300mg, 6 month schedule
- Group 3a: 2 doses of AZD7442 300mg, 10-14 months schedule + 2 doses of AZD7442 600mg, 6 month schedule;
- Group 3b: 1 dose of AZD7442 300mg, 6 month schedule + 2 doses of AZD7442 600mg, 6 month schedule
Period: Provent Main Study
Arm/Group | AZD7442 | Placebo | Group1 | Group 2 | Group 3a | Group 3b
Started (Participants entering the Main Study) | 3460 | 1737 | 0 (This group is for Sub Study only) | 0 (This group is for Sub Study only) | 0 (This group is for Sub Study only) | 0 (This group is for Sub Study only)
Completed (Participants entering the Main Study) | 2490 | 1179 | 0 | 0 | 0 | 0
Not Completed | 970 | 558 | 0 | 0 | 0 | 0
Not completed — PARTICIPANT NOT FULFILLING INCLUSION CRITERIA | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 242 | 144 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 5 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 357 | 200 | 0 | 0 | 0 | 0
Not completed — Death | 22 | 10 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Participants dosed in sub-study | 310 | 193 | 0 | 0 | 0 | 0
Not completed — PARTICIPANT NOT COMPLIANT | 1 | 1 | 0 | 0 | 0 | 0
Not completed — PARTICIPANT COULD NOT BE REACHED PRIOR TO DBL | 14 | 2 | 0 | 0 | 0 | 0
Not completed — INCARCERATION | 3 | 0 | 0 | 0 | 0 | 0
Not completed — WITHDRAWAL OF CONSENT | 3 | 2 | 0 | 0 | 0 | 0
Not completed — MOVED ABROAD / LOCATION | 7 | 2 | 0 | 0 | 0 | 0
Not completed — PARTICIPANT DID NOT ATTEND VISIT | 2 | 2 | 0 | 0 | 0 | 0
Not completed — MISSING REASON | 0 | 1 | 0 | 0 | 0 | 0
Period: Provent Sub Study
Arm/Group | AZD7442 | Placebo | Group1 | Group 2 | Group 3a | Group 3b
Started (Participants in the Sub Study) | 0 (This group is for Main Study only) | 0 (This group is for Main Study only) | 234 | 119 | 76 | 74
Completed (Participants in the Sub Study) | 0 | 0 | 194 | 90 | 64 | 61
Not Completed | 0 | 0 | 40 | 29 | 12 | 13
Not completed — SUBJECT MOVED OUT OF AREA | 0 | 0 | 0 | 1 | 0 | 0
Not completed — SUBJECT WAS MOVING AWAY FROM THE STUDY CLINIC | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 20 | 10 | 6 | 4
Not completed — Death | 0 | 0 | 8 | 5 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1
Not completed — DUE TO SUBJECT'S DECLINING HEALTH THE SUBJECT WILL NO LONGER BE ABLE TO PARTICIPATE IN THE STUDY | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 11 | 13 | 5 | 6
Not completed — NON COMPLIANCE BY SUBJECT | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: This study is made of two parts: Main study (overall number of participants is 5197) and a Sub Study where 503 participants from the Main study took different treatments from Main Study. Total across groups is not applicable here.
Groups:
- Group 1: 2 doses of AZD7442 300mg, 10-14 months schedule
- Group 3a: 2 doses of AZD7442 300mg, 10-14 months schedule + 2 doses of AZD7442 600mg, 6 month schedule
- Total: Total of all reporting groups
Arm/Group | AZD7442 | Placebo | Group 1 | Group 2 | Group 3a | Group 3b | Total
Number analyzed (Participants) | 3460 | 1737 | 234 | 119 | 76 | 74 | 5700
Age, Continuous [Mean (Standard Deviation); unit: Years] — Main Study: FAS population - Sub Study : As Treated Population: This study is made of two parts: Main study (overall number of participants is 5197) and a Sub Study where 503 participants from the Main study were allocated to different treatments with respect to the Main Study. Total across groups is not applicable.
  Years
    Main Study: number analyzed (Participants) | 3460 | 1737 | 0 | 0 | 0 | 0 | 5197
    Main Study | 53.65 (14.99) | 53.27 (14.93) |  |  |  |  | 53.52 (14.97)
    Sub Study: number analyzed (Participants) | 0 | 0 | 234 | 119 | 76 | 74 | 503
    Sub Study |  |  | 60.73 (11.63) | 60.62 (11.56) | 59.29 (11.61) | 59.00 (11.39) | 60.23 (11.56)
Age, Continuous [Median (Full Range); unit: Years] — Main Study: FAS population - Sub Study : As Treated Population: This study is made of two parts: Main study (overall number of participants is 5197) and a Sub Study where 503 participants from the Main study were allocated to different treatments with respect to the Main Study. Total across groups is not applicable.
  Years
    Main Study: number analyzed (Participants) | 3460 | 1737 | 0 | 0 | 0 | 0 | 5197
    Main Study | 57 [18 to 98] | 57 [18 to 99] |  |  |  |  | 57 [18 to 99]
    Sub Study: number analyzed (Participants) | 0 | 0 | 234 | 119 | 76 | 74 | 503
    Sub Study |  |  | 62.0 [21 to 84] | 62.0 [23 to 82] | 60.5 [22 to 86] | 61 [30 to 92] | 62 [21 to 92]
Age, Customized [Count of Participants; unit: Participants] — Main Study: FAS population - Sub Study : As Treated Population: This study is made of two parts: Main study (overall number of participants is 5197) and a Sub Study where 503 participants from the Main study were allocated to different treatments with respect to the Main Study. Total across groups is not applicable.
  Participants
    Main Study : >= 18 - < 60 years: number analyzed (Participants) | 3460 | 1737 | 0 | 0 | 0 | 0 | 5197
    Main Study : >= 18 - < 60 years | 1960 | 980 |  |  |  |  | 2940
    Main Study : >= 60 - < 70 years: number analyzed (Participants) | 3460 | 1737 | 0 | 0 | 0 | 0 | 5197
    Main Study : >= 60 - < 70 years | 1083 | 563 |  |  |  |  | 1646
    Main Study : >= 70 - < 80 years: number analyzed (Participants) | 3460 | 1737 | 0 | 0 | 0 | 0 | 5197
    Main Study : >= 70 - < 80 years | 368 | 174 |  |  |  |  | 542
    Main Study : >= 80 years: number analyzed (Participants) | 3460 | 1737 | 0 | 0 | 0 | 0 | 5197
    Main Study : >= 80 years | 49 | 20 |  |  |  |  | 69
    Sub Study : >= 18 - < 60 years: number analyzed (Participants) | 0 | 0 | 234 | 119 | 76 | 74 | 503
    Sub Study : >= 18 - < 60 years |  |  | 82 | 37 | 31 | 33 | 183
    Sub Study : >= 60 - < 70 years: number analyzed (Participants) | 0 | 0 | 234 | 119 | 76 | 74 | 503
    Sub Study : >= 60 - < 70 years |  |  | 103 | 58 | 33 | 30 | 224
    Sub Study : >= 70 - < 80 years: number analyzed (Participants) | 0 | 0 | 234 | 119 | 76 | 74 | 503
    Sub Study : >= 70 - < 80 years |  |  | 44 | 21 | 8 | 10 | 83
    Sub Study : >= 80 years: number analyzed (Participants) | 0 | 0 | 234 | 119 | 76 | 74 | 503
    Sub Study : >= 80 years |  |  | 5 | 3 | 4 | 1 | 13
Sex: Female, Male [Count of Participants; unit: Participants] — Main Study: FAS population - Sub Study : As Treated Population: This study is made of two parts: Main study (overall number of participants is 5197) and a Sub Study where 503 participants from the Main study were allocated to different treatments with respect to the Main Study. Total across groups is not applicable.
  Participants
    Main Study: number analyzed (Participants) | 3460 | 1737 | 0 | 0 | 0 | 0 | 5197
    Main Study: Female | 1594 | 802 |  |  |  |  | 2396
    Main Study: Male | 1866 | 935 |  |  |  |  | 2801
    Sub Study: number analyzed (Participants) | 0 | 0 | 234 | 119 | 76 | 74 | 503
    Sub Study: Female |  |  | 113 | 48 | 33 | 35 | 229
    Sub Study: Male |  |  | 121 | 71 | 43 | 39 | 274
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Main Study: FAS population - Sub Study : As Treated Population: This study is made of two parts: Main study (overall number of participants is 5197) and a Sub Study where 503 participants from the Main study were allocated to different treatments with respect to the Main Study. Total across groups is not applicable.
  Participants
    Main Study: number analyzed (Participants) | 3460 | 1737 | 0 | 0 | 0 | 0 | 5197
    Main Study: Hispanic or Latino | 539 | 215 |  |  |  |  | 754
    Main Study: Not Hispanic or Latino | 2731 | 1412 |  |  |  |  | 4143
    Main Study: Not reported | 116 | 72 |  |  |  |  | 188
    Main Study: Unknown | 74 | 38 |  |  |  |  | 112
    Sub Study: number analyzed (Participants) | 0 | 0 | 234 | 119 | 76 | 74 | 503
    Sub Study: Hispanic or Latino |  |  | 31 | 6 | 9 | 12 | 58
    Sub Study: Not Hispanic or Latino |  |  | 192 | 109 | 61 | 56 | 418
    Sub Study: Not reported |  |  | 9 | 3 | 4 | 4 | 20
    Sub Study: Unknown |  |  | 2 | 1 | 2 | 2 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Main Study: FAS population - Sub Study : As Treated Population: This study is made of two parts: Main study (overall number of participants is 5197) and a Sub Study where 503 participants from the Main study were allocated to different treatments with respect to the Main Study. Total across groups is not applicable
  Participants
    Main Study: number analyzed (Participants) | 3460 | 1737 | 0 | 0 | 0 | 0 | 5197
    Main Study: White | 2545 | 1249 |  |  |  |  | 3794
    Main Study: Black or African American | 597 | 302 |  |  |  |  | 899
    Main Study: Asian | 110 | 60 |  |  |  |  | 170
    Main Study: American Indian or Alaska Native | 19 | 10 |  |  |  |  | 29
    Main Study: Native Hawaiian or Other Pacific Islander | 4 | 4 |  |  |  |  | 8
    Main Study: Not reported | 89 | 56 |  |  |  |  | 145
    Main Study: Unknown | 79 | 42 |  |  |  |  | 121
    Main Study: Other | 15 | 12 |  |  |  |  | 27
    Main Study: Missing | 2 | 2 |  |  |  |  | 4
    Sub Study: number analyzed (Participants) | 0 | 0 | 234 | 119 | 76 | 74 | 503
    Sub Study: White |  |  | 204 | 106 | 52 | 53 | 415
    Sub Study: Black or African American |  |  | 20 | 11 | 14 | 14 | 59
    Sub Study: Asian |  |  | 4 | 1 | 6 | 1 | 12
    Sub Study: American Indian or Alaska Native |  |  | 0 | 0 | 0 | 0 | 0
    Sub Study: Native Hawaiian or Other Pacific Islander |  |  | 0 | 0 | 0 | 0 | 0
    Sub Study: Not reported |  |  | 2 | 0 | 0 | 1 | 3
    Sub Study: Unknown |  |  | 4 | 1 | 4 | 3 | 12
    Sub Study: Other |  |  | 0 | 0 | 0 | 2 | 2
    Sub Study: Missing |  |  | 0 | 0 | 0 | 0 | 0
SARS-CoV-2 status at baseline [Count of Participants; unit: Participants] — Main Study: FAS population - Sub Study : As Treated Population: This study is made of two parts: Main study (overall number of participants is 5197) and a Sub Study where 503 participants from the Main study were allocated to different treatments with respect to the Main Study. Total across groups is not applicable
  Participants
    Main Study: number analyzed (Participants) | 3460 | 1737 | 0 | 0 | 0 | 0 | 5197
    Main Study: Positive | 19 | 6 |  |  |  |  | 25
    Main Study: Negative | 3316 | 1665 |  |  |  |  | 4981
    Main Study: Missing | 125 | 66 |  |  |  |  | 191
    Sub Study: number analyzed (Participants) | 0 | 0 | 234 | 119 | 76 | 74 | 503
    Sub Study: Positive |  |  | 0 | 1 | 0 | 1 | 2
    Sub Study: Negative |  |  | 229 | 114 | 75 | 70 | 488
    Sub Study: Missing |  |  | 5 | 4 | 1 | 3 | 13
Region [Count of Participants; unit: Participants] — Main Study: FAS population - Sub Study : As Treated Population: This study is made of two parts: Main study (overall number of participants is 5197) and a Sub Study where 503 participants from the Main study were allocated to different treatments with respect to the Main Study. Total across groups is not applicable
  Participants
    Main Study: number analyzed (Participants) | 3460 | 1737 | 0 | 0 | 0 | 0 | 5197
    Main Study: North America | 2487 | 1232 |  |  |  |  | 3719
    Main Study: United Kingdom | 611 | 312 |  |  |  |  | 923
    Main Study: European Union | 362 | 193 |  |  |  |  | 555
    Sub Study: number analyzed (Participants) | 0 | 0 | 234 | 119 | 76 | 74 | 503
    Sub Study: North America |  |  | 130 | 75 | 76 | 74 | 355
    Sub Study: United Kingdom |  |  | 77 | 27 | 0 | 0 | 104
    Sub Study: European Union |  |  | 27 | 17 | 0 | 0 | 44
Any COVID-19 comorbidities at baseline [Count of Participants; unit: Participants] — Main Study: FAS population - Sub Study : As Treated Population: This study is made of two parts: Main study (overall number of participants is 5197) and a Sub Study where 503 participants from the Main study were allocated to different treatments with respect to the Main Study. Total across groups is not applicable
  Participants
    Main Study: number analyzed (Participants) | 3460 | 1737 | 0 | 0 | 0 | 0 | 5197
    Main Study: Yes | 2432 | 1206 |  |  |  |  | 3638
    Main Study: Missing | 1028 | 531 |  |  |  |  | 1559
    Sub Study: number analyzed (Participants) | 0 | 0 | 234 | 119 | 76 | 74 | 503
    Sub Study: Yes |  |  | 192 | 97 | 66 | 68 | 423
    Sub Study: Missing |  |  | 42 | 22 | 10 | 6 | 80
Any high risk for severe COVID-19 at baseline [Count of Participants; unit: Participants] — Main Study: FAS population - Sub Study : As Treated Population: This study is made of two parts: Main study (overall number of participants is 5197) and a Sub Study where 503 participants from the Main study were allocated to different treatments with respect to the Main Study. Total across groups is not applicable
  Participants
    Main Study: number analyzed (Participants) | 3460 | 1737 | 0 | 0 | 0 | 0 | 5197
    Main Study: Yes | 2674 | 1366 |  |  |  |  | 4040
    Main Study: Missing | 786 | 371 |  |  |  |  | 1157
    Sub Study: number analyzed (Participants) | 0 | 0 | 234 | 119 | 76 | 74 | 503
    Sub Study: Yes |  |  | 209 | 107 | 69 | 73 | 458
    Sub Study: Missing |  |  | 25 | 12 | 7 | 1 | 45
Height [Mean (Standard Deviation); unit: cm] — Main Study: FAS population - Sub Study : As Treated Population: This study is made of two parts: Main study (overall number of participants is 5197) and a Sub Study where 503 participants from the Main study were allocated to different treatments with respect to the Main Study. Total across groups is not applicable
  cm
    Main Study: number analyzed (Participants) | 3460 | 1737 | 0 | 0 | 0 | 0 | 5197
    Main Study | 170.04 (10.10) | 170.17 (9.84) |  |  |  |  | 170.9 (10.02)
    Sub Study: number analyzed (Participants) | 0 | 0 | 234 | 119 | 76 | 74 | 503
    Sub Study |  |  | 170.03 (10.29) | 171.25 (10.06) | 169.03 (9.76) | 168.72 (10.27) | 169.97 (10.16)
Baseline BMI [Mean (Standard Deviation); unit: kg/m**2] — Main Study: FAS population - Sub Study : As Treated Population: This study is made of two parts: Main study (overall number of participants is 5197) and a Sub Study where 503 participants from the Main study were allocated to different treatments with respect to the Main Study. Total across groups is not applicable
  kg/m**2
    Main Study: number analyzed (Participants) | 3460 | 1737 | 0 | 0 | 0 | 0 | 5197
    Main Study | 29.57 (6.88) | 29.62 (6.98) |  |  |  |  | 29.59 (6.91)
    Sub Study: number analyzed (Participants) | 0 | 0 | 234 | 119 | 76 | 74 | 503
    Sub Study |  |  | 29.72 (6.00) | 28.88 (6.31) | 29.67 (7.06) | 31.50 (7.06) | 29.78 (6.43)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With First Case of SARS-CoV-2 RT-PCR-positive Symptomatic Illness
Description: To estimate the efficacy of a single IM dose of AZD7442 compared to placebo for the prevention of COVID-19 prior to Day 183. Planned to be evaluated through Day 183, however, the number of events required for the primary endpoint was achieved 165 days after the study start date which is displayed in the primary efficacy row below. Final analysis is final data from the study based on the pre-planned 183 days of follow up for this endpoint.
Time Frame: 165 Days for primary analysis, 183 days for final analysis
Population: All randomized and dosed participants who did not have a prior SARS-CoV-2 RT-PCR-positive confirmed COVID-19 infection.
Measure: Count of Participants; unit: Participants
Arm/Group | AZD7442 | Placebo
Number analyzed (Participants) | 3441 | 1731
Participants
  Primary Analysis | 8 | 17
  Final Analysis | 12 | 34
Statistical Analysis 1: Comparison: AZD7442 vs Placebo; Primary Analysis; Test type: Superiority; p < 0.001, Poisson regression; Relative Risk Reduction = 76.73, 95% CI 2-sided [46.05 to 89.96] — Estimates are based on a Poisson regression with robust variance. The model includes covariate for treatment, and age group, with the log of the follow-up time as an offset. Estimated RRR greater than 0% provides evidence in favor of AZD7442
Statistical Analysis 2: Comparison: AZD7442 vs Placebo; Final Analysis; Test type: Superiority; p < 0.001, Poisson regression; Relative Risk Reduction = 83.04, 95% CI 2-sided [67.26 to 91.21] — [estimate comment as in outcome 1, analysis 1]

2. Other Pre Specified Outcome: AEs, SAEs, MAAEs, and AESIs Post Dose of IMP at Time of Primary Efficacy Analysis
Description: To assess the safety and tolerability of a single IM dose of AZD7442 compared to placebo
Time Frame: 165 Days
Population: All participants dosed
Measure: Count of Participants; unit: Participants
Arm/Group | AZD7442 | Placebo
Number analyzed (Participants) | 3461 | 1736
Participants
  Adverse Events | 1221 | 593
  Serious Adverse Events | 50 | 23
  Medically Attended Adverse Events | 360 | 157
  Adverse Events of Special Interest | 93 | 37

3. Secondary Outcome: The Incidence of Participants Who Have a Post-treatment Response (Negative at Baseline to Positive at Any Time Post-baseline) for SARS-CoV-2 Nucleocapsid Antibodies.
Description: To estimate the efficacy of a single IM dose of AZD7442 compared to placebo for the prevention of SARS-CoV-2 infection
Time Frame: 366 days
Population: All randomized and dosed participants who did not have a prior SARS-CoV-2 RT-PCR-positive confirmed COVID-19 infection and had an evaluable sample obtained.
Measure: Count of Participants; unit: Participants
Arm/Group | AZD7442 | Placebo
Number analyzed (Participants) | 3121 | 1563
Participants | 198 | 139
Statistical Analysis 1: Comparison: AZD7442 vs Placebo; Test type: Superiority; p < 0.001, Poisson regression; Relative Risk Reduction = 34.90, 95% CI 2-sided [21.44 to 46.05] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: The Incidence of SARS-CoV-2 RT-PCR-positive Severe or Critical Symptomatic Illness Occurring After Dosing With IMP
Description: To estimate the efficacy of a single IM dose of AZD7442 compared to placebo for the prevention of severe or critical symptomatic COVID-19
Time Frame: 366 Days
Population: All randomized and dosed participants who did not have a prior SARS-CoV-2 RT-PCR-positive confirmed COVID-19 infection
Measure: Count of Participants; unit: Participants
Arm/Group | AZD7442 | Placebo
Number analyzed (Participants) | 3441 | 1731
Participants | 2 | 11
Statistical Analysis 1: Comparison: AZD7442 vs Placebo; Test type: Superiority; p = 0.001, Poisson regression; Relative Risk Reduction = 91.41, 95% CI 2-sided [61.31 to 98.09] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: The Incidence of COVID-19-related Emergency Department Visits Occurring After Dosing With IMP
Description: To estimate the efficacy of a single IM dose of AZD7442 compared to placebo for the prevention of COVID-19-related Emergency Department visits
Time Frame: 366 days
Population: All randomized and dosed participants who did not have a prior SARS-CoV-2 RT-PCR-positive confirmed COVID-19 infection
Measure: Count of Participants; unit: Participants
Arm/Group | AZD7442 | Placebo
Number analyzed (Participants) | 3441 | 1731
Participants | 8 | 8
Statistical Analysis 1: Comparison: AZD7442 vs Placebo; Test type: Superiority; p = 0.137, Poisson regression; Relative Risk Reduction = 52.43, 95% CI 2-sided [-26.61 to 82.13]

6. Secondary Outcome: Serum AZD7442 Concentrations, PK Parameters if Data Permit.
Description: To assess the pharmacokinetics of AZD7442 administered as a single dose of 300 mg IM
Time Frame: 457 days
Population: PK analysis set (only AZD7442 arm)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | AZD7442 | Placebo
Number analyzed (Participants) | 3290 | 0
µg/mL
  Day 8: number analyzed (Participants) | 3155 | 0
  Day 8 | 18.667 (92.947) |
  Day 29: number analyzed (Participants) | 3106 | 0
  Day 29 | 22.602 (64.691) |
  Day 58: number analyzed (Participants) | 3103 | 0
  Day 58 | 18.707 (65.981) |
  Day 92: number analyzed (Participants) | 3008 | 0
  Day 92 | 14.037 (67.922) |
  Day 183: number analyzed (Participants) | 2969 | 0
  Day 183 | 5.593 (83.580) |
  Day 366: number analyzed (Participants) | 2691 | 0
  Day 366 | 1.340 (90.132) |
  Day 457: number analyzed (Participants) | 1963 | 0
  Day 457 | 0.565 (85.733) |

7. Secondary Outcome: Incidence of ADA to AZD7442 in Serum
Description: To evaluate ADA responses to AZD7442 in serum
Time Frame: 457 days
Population: AZD7442 ADA Evaluable Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | AZD7442 | Placebo
Number analyzed (Participants) | 3086 | 1540
Participants | 403 | 34

8. Primary Outcome: AEs, SAEs, MAAEs, and AESIs Post Dose of IMP
Description: To assess the safety and tolerability of a single IM dose of AZD7442 compared to placebo
Time Frame: 457 Days, Final analysis
Population: All participants dosed
Measure: Count of Participants; unit: Participants
Arm/Group | AZD7442 | Placebo
Number analyzed (Participants) | 3461 | 1736
Participants
  Adverse Events | 2016 | 1007
  Serious Adverse Events | 215 | 97
  Medically Attended Adverse Events | 991 | 439
  Adverse Events of Special Interest | 103 | 43

ADVERSE EVENTS:
Time Frame: All AEs were collected from the time of IMP administration throughout the study, up to and including the last visit. For the Main study the duration of follow up from Dose of IMP to End of Study (Days) was in the range of 1-605. For the Sub Study the range was 1-688 days.
Groups:
- AZD7442; Placebo; Group 1; Group 2; Group 3a; Group 3b: Description (Arm-group)
Arm/Group | AZD7442 | Placebo | Group 1 | Group 2 | Group 3a | Group 3b
All-Cause Mortality (participants affected / at risk) | 22/3461 | 10/1736 | 8/234 | 5/119 | 0/76 | 1/74
Serious Adverse Events (participants affected / at risk) | 215/3461 | 97/1736 | 31/234 | 20/119 | 12/76 | 12/74
Other Adverse Events (participants affected / at risk) | 1988/3461 | 993/1736 | 185/234 | 94/119 | 58/76 | 55/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD7442 (N=3461) | Placebo (N=1736) | Group 1 (N=234) | Group 2 (N=119) | Group 3a (N=76) | Group 3b (N=74)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adrenal gland cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervix carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon cancer stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
External ear neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung adenocarcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung adenocarcinoma stage iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papillary renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bell's palsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carotid artery disease (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral venous sinus thrombosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Inner ear disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Complex regional pain syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dementia alzheimer's type (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lacunar infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ruptured cerebral aneurysm (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Simple partial seizures (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thalamic infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device deposit issue (Product Issues) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Psychiatric decompensation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 5 (5) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvi-ureteric obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subcapsular renal haematoma (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Thyrotoxic crisis (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 3 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sexual abuse (Social circumstances) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Withdrawal of life support (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertensive urgency (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Secondary hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterovesical fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gallstone ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intra-abdominal fluid collection (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mesenteric artery thrombosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Overflow diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis relapsing (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritoneal cyst (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Salivary gland mass (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Volvulus (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 8 (8) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 4 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gallbladder obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis perforated (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriovenous graft site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 2 (2) | 6 (6) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Covid-19 pneumonia (Infections and infestations) | 4 (4) | 20 (20) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Campylobacter infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 6 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3)
Enterococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Extradural abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gangrene (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis e (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incision site cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meningitis streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 6 (6) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 7 (8) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
Cardiomegaly (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia fungal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Secondary syphilis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 7 (7) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Sialoadenitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vestibular neuronitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral diarrhoea (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Incisional hernia, obstructive (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mitral valve disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritoneal dialysis complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Second degree chemical burn of skin (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 7 (7) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sternal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paroxysmal atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcoholic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes with hyperosmolarity (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint instability (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD7442 (N=3461) | Placebo (N=1736) | Group 1 (N=234) | Group 2 (N=119) | Group 3a (N=76) | Group 3b (N=74)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 17 (17) | 6 (6) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 11 (14) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 185 (207) | 90 (102) | 28 (34) | 20 (25) | 6 (7) | 2 (2)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 12 (12) | 12 (12) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 35 (37) | 20 (21) | 7 (7) | 3 (4) | 1 (1) | 1 (1)
Thalassaemia beta (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 8 (8) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 45 (49) | 25 (27) | 5 (5) | 0 (0) | 1 (1) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Type v hyperlipidaemia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 7 (10) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 3 (3) | 9 (9) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scapholunate dissociation (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 6 (9) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Soft tissue mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 10 (11) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spondylitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendon calcification (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 2 (4) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 6 (7) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal wall neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deafness bilateral (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 5 (6) | 5 (6) | 2 (2) | 0 (0) | 0 (0)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blepharal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer fatigue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deafness unilateral (Ear and labyrinth disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysplastic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Essential thrombocythaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear canal erythema (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eyelid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemangioma of bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hair follicle tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypergammaglobulinaemia benign monoclonal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear congestion (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant neoplasm of eyelid (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myeloproliferative neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hilar lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 13 (13) | 9 (9) | 1 (1) | 1 (2) | 1 (1) | 0 (0)
Naevus haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Plasma cell myeloma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 3 (3) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Excessive cerumen production (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tongue neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ageusia (Nervous system disorders) | 63 (67) | 35 (37) | 8 (8) | 5 (6) | 1 (1) | 3 (3)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
External ear inflammation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anosmia (Nervous system disorders) | 57 (60) | 30 (31) | 7 (8) | 5 (7) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Axonal neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bell's palsy (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burning sensation (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carotid arteriosclerosis (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Haematotympanum (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carotid artery occlusion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Carotid artery thrombosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Central pain syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral arteriosclerosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral artery occlusion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral atrophy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral congestion (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral microangiopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral small vessel ischaemic disease (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervicogenic headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic inflammatory demyelinating polyradiculoneuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clonus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cluster headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 3 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Complex regional pain syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cranial nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cubital tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dementia (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inner ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 52 (56) | 22 (28) | 5 (5) | 3 (5) | 1 (1) | 3 (3)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 3 (4) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Essential tremor (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial paresis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Middle ear effusion (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fine motor skill dysfunction (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head discomfort (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 439 (564) | 211 (252) | 52 (64) | 33 (42) | 7 (11) | 8 (9)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersomnia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 13 (13) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otorrhoea (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypogeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyposmia (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intercostal neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intraneural cyst (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 7 (7) | 5 (5) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Leukoencephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperleukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presbyacusis (Ear and labyrinth disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental impairment (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 24 (27) | 8 (10) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Migraine with aura (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Movement disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle contractions involuntary (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myelopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myoclonus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sudden hearing loss (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nerve compression (Nervous system disorders) | 3 (3) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 3 (3) | 7 (7) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Normal pressure hydrocephalus (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ophthalmic migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osmotic demyelination syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 17 (17) | 10 (10) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Parkinson's disease (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parosmia (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral nerve lesion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Superior semicircular canal dehiscence (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peroneal nerve palsy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Piriformis syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Psychomotor hyperactivity (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radicular pain (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radiculopathy (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 7 (7) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 16 (17) | 7 (8) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 5 (6) | 3 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus headache (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Speech disorder (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Spinal claudication (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 16 (17) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Taste disorder (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient global amnesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 6 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Trigeminal neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular dementia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage in pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 17 (20) | 7 (9) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Device breakage (Product Issues) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device loosening (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device malfunction (Product Issues) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device occlusion (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device physical property issue (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute stress disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aggression (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 5 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alcoholism (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anger (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 34 (36) | 11 (11) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Anxiety disorder (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Autism spectrum disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Borderline personality disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Claustrophobia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Addison's disease (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 15 (15) | 9 (9) | 4 (5) | 2 (2) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 7 (7) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 22 (22) | 8 (8) | 2 (2) | 3 (3) | 0 (0) | 3 (3)
Disorientation (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug abuse (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug use disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Euphoric mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalised anxiety disorder (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Grief reaction (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adrenomegaly (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hallucinations, mixed (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 21 (22) | 14 (14) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mania (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mixed anxiety and depressive disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervousness (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nightmare (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obsessive-compulsive disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Androgen deficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Panic disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Persistent complex bereavement disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rapid eye movement sleep behaviour disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 7 (7) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sleep terror (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somatic symptom disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Autoimmune thyroiditis (Endocrine disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 5 (5) | 10 (11) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Bladder cyst (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder outlet obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chromaturia (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 7 (7) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (3)
Crystalluria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 9 (9) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glycosuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 22 (23) | 10 (10) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Haemorrhage urinary tract (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Leukocyturia (Renal and urinary disorders) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lupus nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Microalbuminuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Micturition disorder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 13 (13) | 8 (9) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Nocturia (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 4 (4) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 6 (7) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal cyst (Renal and urinary disorders) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stag horn calculus (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress urinary incontinence (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urethral meatus stenosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urge incontinence (Renal and urinary disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 4 (4) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypogonadism (Endocrine disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal uterine bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenomyosis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Balanoposthitis (Reproductive system and breast disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bartholin's cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 9 (9) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Breast calcifications (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cyst (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast enlargement (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast mass (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothalamo-pituitary disorder (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast swelling (Reproductive system and breast disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervix inflammation (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ejaculation failure (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epididymal cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibrocystic breast disease (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 9 (9) | 5 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Menometrorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Menopausal disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Menopausal symptoms (Reproductive system and breast disorders) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nipple pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oligomenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pituitary cyst (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic adhesions (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic congestion (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Perineal pain (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peyronie's disease (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polycystic ovaries (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Premenstrual syndrome (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Priapism (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Primary hypogonadism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Testicular cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urogenital atrophy (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal prolapse (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varicocele (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thyroid atrophy (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulva cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal inflammation (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Allergic bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 19 (22) | 8 (9) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroid mass (Endocrine disorders) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Asthma exercise induced (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 19 (22) | 8 (14) | 4 (4) | 2 (3) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 423 (517) | 179 (213) | 68 (88) | 36 (58) | 14 (21) | 10 (10)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 4 (4) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 162 (225) | 67 (92) | 26 (43) | 18 (29) | 5 (7) | 4 (6)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 6 (6) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Age-related macular degeneration (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal leukoplakia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal cavity mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 283 (320) | 114 (128) | 42 (52) | 26 (34) | 11 (11) | 8 (9)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal pruritus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 305 (357) | 117 (135) | 47 (56) | 21 (34) | 9 (12) | 7 (9)
Astigmatism (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal plaque (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 19 (19) | 9 (10) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Pulmonary artery dilatation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 25 (26) | 8 (8) | 0 (0) | 3 (4) | 2 (2) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 2 (3) | 1 (1) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 11 (12) | 5 (5) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Reflux laryngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory gas exchange disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chalazion (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 316 (363) | 124 (141) | 43 (54) | 29 (40) | 8 (14) | 6 (6)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinonasal obstruction (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 38 (45) | 15 (20) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 21 (24) | 11 (11) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suffocation feeling (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 4 (4) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsillar erythema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tracheal disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vasomotor rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 15 (16) | 9 (9) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 7 (7) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 7 (7) | 3 (3) | 2 (2) | 4 (5) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 5 (5) | 4 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 6 (6) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 3 (3) | 2 (2) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 10 (10) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (2)
Diabetic wound (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 7 (7) | 3 (5) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 7 (7) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dacryostenosis acquired (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Granuloma annulare (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hidradenitis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hirsutism (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 7 (7) | 5 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkeratosis follicularis et parafollicularis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intertrigo (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lichen sclerosus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatochalasis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipodystrophy acquired (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Macule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 11 (12) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Penile ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photodermatosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic retinal oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 21 (21) | 13 (13) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Pruritus allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Purpura senile (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 41 (46) | 22 (22) | 0 (0) | 3 (4) | 2 (3) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic retinopathy (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sensitive skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 4 (5) | 8 (9) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Skin oedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin plaque (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin striae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry age-related macular degeneration (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 11 (12) | 5 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alcohol use (Social circumstances) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Menopause (Social circumstances) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Physical abuse (Social circumstances) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Physical assault (Social circumstances) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angiodysplasia (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 9 (9) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Aortic dilatation (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arteriovenous fistula (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure fluctuation (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood pressure inadequately controlled (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 8 (9) | 3 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Essential hypertension (Vascular disorders) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema of eyelid (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 10 (10) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 99 (102) | 56 (60) | 12 (12) | 7 (9) | 8 (9) | 6 (6)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertensive emergency (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertensive urgency (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 10 (10) | 5 (5) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Intermittent claudication (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye allergy (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurogenic shock (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral venous disease (Vascular disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Raynaud's phenomenon (Vascular disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subclavian vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye inflammation (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Varicose vein (Vascular disorders) | 6 (6) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vascular pain (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White coat hypertension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 5 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 4 (4) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye swelling (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 3 (3) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 5 (6) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Macular degeneration (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Macular fibrosis (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Macular oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular hypertension (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ophthalmoplegia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Orbital oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital oedema (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital swelling (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Posterior capsule opacification (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presbyopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pterygium (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Retinal tear (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scleritis (Eye disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling of eyelid (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uveitis (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual field defect (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vitreous adhesions (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitreous detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 9 (9) | 7 (8) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal mass (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 29 (30) | 19 (21) | 7 (7) | 4 (5) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 11 (11) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 21 (22) | 7 (7) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 37 (37) | 17 (17) | 1 (1) | 3 (3) | 1 (2) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 15 (18) | 8 (8) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Abdominal rigidity (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal pruritus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal skin tags (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angular cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anogenital dysplasia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anorectal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Apical granuloma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bile acid malabsorption (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bowel movement irregularity (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Change of bowel habit (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coeliac disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 4 (4) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis microscopic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 25 (26) | 11 (12) | 5 (5) | 3 (3) | 1 (1) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 5 (6) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diaphragmatic hernia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 183 (206) | 81 (91) | 23 (26) | 16 (22) | 5 (5) | 3 (3)
Diverticulum (Gastrointestinal disorders) | 11 (11) | 0 (0) | 2 (2) | 3 (3) | 2 (2) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Macrocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 7 (7) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyskinesia oesophageal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 13 (13) | 7 (7) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 7 (7) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Eosinophilic oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faeces soft (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 3 (4) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric disorder (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 10 (10) | 3 (3) | 1 (1) | 0 (0) | 4 (4) | 2 (2)
Gastritis alcoholic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 5 (6) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal hypermotility (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal mucosa hyperaemia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 28 (28) | 14 (15) | 5 (5) | 5 (5) | 1 (1) | 2 (2)
Giant cell epulis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glossitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 4 (4) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 15 (15) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids thrombosed (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 9 (9) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperaesthesia teeth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inflammatory bowel disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia strangulated (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 7 (8) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lip disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Loose tooth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 5 (5) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 163 (191) | 75 (82) | 14 (16) | 8 (12) | 8 (11) | 6 (6)
Odynophagia (Gastrointestinal disorders) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal dilatation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal motility disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal spasm (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Polycythaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral disorder (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral mucosal blistering (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral mucosal eruption (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic failure (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatic mass (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic steatosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Splenomegaly (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Plicated tongue (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 5 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rectal polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Salivary gland disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Salivary gland enlargement (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Salivary gland mucocoele (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sigmoid mesocolon hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Submaxillary gland enlargement (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swollen tongue (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue discolouration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tongue discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue erythema (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tongue geographic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue ulceration (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth impacted (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth loss (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 17 (18) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Trichoglossia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 5 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uvulitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 60 (75) | 30 (33) | 10 (10) | 3 (3) | 2 (3) | 3 (3)
Adverse drug reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 19 (20) | 14 (14) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Axillary pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 9 (10) | 7 (8) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 9 (9) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 155 (169) | 72 (79) | 21 (22) | 17 (22) | 6 (7) | 5 (5)
Chronic fatigue syndrome (General disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Crepitations (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cyst (General disorders) | 3 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug withdrawal syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Energy increased (General disorders) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facial pain (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 369 (439) | 166 (201) | 54 (68) | 33 (49) | 11 (14) | 6 (6)
Feeling abnormal (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Feeling cold (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling jittery (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foaming at mouth (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 3 (3) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hangover (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 10 (10) | 4 (4) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Hernia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inflammation (General disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 27 (29) | 14 (16) | 3 (3) | 4 (11) | 1 (1) | 0 (0)
Injection site bruising (General disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site discomfort (General disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 8 (9) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site haematoma (General disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site haemorrhage (General disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site induration (General disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site joint pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site mass (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site oedema (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 37 (39) | 19 (20) | 1 (1) | 1 (1) | 4 (5) | 0 (0)
Injection site paraesthesia (General disorders) | 3 (3) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 9 (9) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site rash (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 6 (7) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 4 (4) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site urticaria (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site warmth (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic valve sclerosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injury associated with device (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 46 (46) | 10 (10) | 8 (8) | 4 (4) | 1 (1) | 0 (0)
Mass (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device site irritation (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 14 (14) | 6 (6) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Oedema (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 17 (18) | 8 (9) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Pain (General disorders) | 185 (212) | 79 (82) | 25 (30) | 19 (20) | 8 (9) | 5 (5)
Peripheral swelling (General disorders) | 15 (16) | 10 (10) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Puncture site oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Puncture site pruritus (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 150 (158) | 77 (84) | 23 (28) | 15 (17) | 6 (7) | 5 (5)
Retention cyst (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Secretion discharge (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sensation of foreign body (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling face (General disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vaccination site discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaccination site erythema (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaccination site mass (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaccination site pain (General disorders) | 8 (8) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaccination site reaction (General disorders) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site bruise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site haematoma (General disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site haemorrhage (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary dyskinesia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 7 (7) | 5 (5) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic cytolysis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic fibrosis (Hepatobiliary disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 11 (11) | 7 (7) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Hepatobiliary cyst (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatosplenomegaly (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperplastic cholecystopathy (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nonalcoholic fatty liver disease (Hepatobiliary disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial enlargement (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergy to arthropod bite (Immune system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergy to arthropod sting (Immune system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergy to chemicals (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergy to plants (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 6 (6) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypogammaglobulinaemia (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mite allergy (Immune system disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 13 (13) | 6 (6) | 2 (2) | 3 (3) | 3 (3) | 2 (2)
Primary amyloidosis (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sarcoidosis (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 29 (29) | 11 (11) | 4 (5) | 2 (2) | 0 (0) | 1 (1)
Abdominal abscess (Infections and infestations) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Acarodermatitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 9 (9) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal chlamydia infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arteriovenous graft site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asymptomatic covid-19 (Infections and infestations) | 28 (28) | 17 (17) | 9 (9) | 7 (7) | 3 (3) | 1 (1)
Asymptomatic bacteriuria (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial disease carrier (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Bacteriuria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Balanitis candida (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Beta haemolytic streptococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Body tinea (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 32 (35) | 10 (10) | 2 (2) | 2 (3) | 0 (0) | 0 (0)
Bronchitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 465 (475) | 229 (240) | 64 (69) | 35 (39) | 13 (15) | 12 (12)
Covid-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 14 (14) | 6 (6) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Cervicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chlamydial infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Chronic sinusitis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Coccidioidomycosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 4 (4) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis bacterial (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 19 (22) | 7 (7) | 2 (2) | 1 (4) | 0 (0) | 1 (1)
Cystitis escherichia (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dacryocanaliculitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dengue haemorrhagic fever (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatophytosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 9 (11) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 14 (14) | 9 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone marrow oedema (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bifascicular block (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterobiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epididymitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Escherichia infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 4 (4) | 5 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Febrile infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Fungaemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 4 (4) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 6 (6) | 7 (7) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 21 (21) | 10 (10) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 5 (5) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal bacterial overgrowth (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bundle branch block left (Cardiac disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Genitourinary chlamydia infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gingival abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gonococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Gonorrhoea (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hiv peripheral neuropathy (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bundle branch block right (Cardiac disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Haemophilus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Helicobacter infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatitis c (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Herpes simplex reactivation (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 16 (16) | 7 (7) | 4 (4) | 2 (2) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 8 (9) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Impetigo (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infected bite (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected cyst (Infections and infestations) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infected dermal cyst (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected skin ulcer (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infective exacerbation of bronchiectasis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 12 (13) | 5 (6) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral discitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Klebsiella infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Labyrinthitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 5 (6) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 27 (30) | 20 (22) | 7 (9) | 2 (2) | 0 (0) | 0 (0)
Lower respiratory tract infection bacterial (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection viral (Infections and infestations) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lyme disease (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphangitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mastitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mastoiditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device site abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Molluscum contagiosum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucormycosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail bed infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal vestibulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 42 (47) | 26 (26) | 12 (12) | 4 (5) | 0 (0) | 0 (0)
Norovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Onychomycosis (Infections and infestations) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oral candidiasis (Infections and infestations) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Oral fungal infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 14 (14) | 8 (9) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orchitis (Infections and infestations) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal candidiasis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal gonococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 8 (9) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 3 (3) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Otitis media acute (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papilloma viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parotitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic inflammatory disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Perichondritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periodontitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pertussis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 17 (18) | 12 (13) | 2 (2) | 3 (4) | 0 (0) | 0 (0)
Pharyngitis bacterial (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 4 (4) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pilonidal cyst (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 21 (22) | 4 (4) | 3 (3) | 1 (1) | 2 (2) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiomegaly (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post-acute covid-19 syndrome (Infections and infestations) | 1 (1) | 2 (4) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proctitis gonococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pustule (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyuria (Infections and infestations) | 9 (10) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Respiratory tract chlamydial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 5 (5) | 6 (6) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 34 (37) | 15 (18) | 2 (4) | 3 (3) | 0 (0) | 0 (0)
Chronotropic incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Root canal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Secondary syphilis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sialoadenitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 34 (39) | 19 (23) | 8 (9) | 3 (3) | 2 (2) | 1 (1)
Sinusitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sinusitis fungal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin bacterial infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 7 (7) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 6 (6) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Spirochaetal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suspected covid-19 (Infections and infestations) | 4 (5) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syphilis (Infections and infestations) | 6 (6) | 5 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Systemic candida (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinea cruris (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinea versicolour (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 8 (8) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 14 (14) | 5 (5) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 15 (15) | 6 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Trichomoniasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 54 (59) | 34 (44) | 8 (9) | 8 (8) | 2 (3) | 2 (3)
Upper respiratory tract infection bacterial (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urethritis gonococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 122 (146) | 59 (63) | 13 (13) | 10 (16) | 6 (7) | 6 (6)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral diarrhoea (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 21 (23) | 12 (12) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Diastolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral rhinitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 15 (15) | 7 (7) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 3 (3) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accident at work (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 2 (2) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Anaesthetic complication (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 9 (10) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Avulsion fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Barotitis media (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cartilage injury (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chemical burns of eye (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Complications of transplant surgery (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 3 (3) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 22 (24) | 4 (4) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Corneal abrasion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epicondylitis (Injury, poisoning and procedural complications) | 6 (6) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Extradural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left atrial enlargement (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 44 (44) | 17 (17) | 9 (9) | 7 (7) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 15 (15) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foreign body (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foreign body in ear (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foreign body in eye (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Graft complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemodialysis complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 4 (4) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 10 (10) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Heat exhaustion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyphaema (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection related reaction (Injury, poisoning and procedural complications) | 10 (13) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 3 (3) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 6 (6) | 8 (8) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Ligament injury (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 18 (18) | 6 (6) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 11 (11) | 9 (9) | 3 (3) | 2 (2) | 0 (0) | 1 (1)
Lip injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left ventricular hypertrophy (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Median nerve injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 4 (4) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle rupture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 8 (8) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Neck injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nerve injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteochondral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic bone injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post concussion syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural constipation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural diarrhoea (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Postoperative delirium (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 10 (11) | 10 (11) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 4 (4) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 6 (6) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Mitral valve stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Second degree chemical burn of skin (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 8 (10) | 4 (4) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Skin injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 22 (25) | 7 (7) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal column injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Splinter (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stab wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomal hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Traumatic ulcer (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ulnar nerve injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 71 (132) | 50 (81) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 8 (8) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anti factor viii antibody increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aortic bruit (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 6 (6) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacterial test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 17 (21) | 10 (10) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Blood hiv rna increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood calcium increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 9 (9) | 3 (3) | 5 (5) | 2 (2) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 24 (24) | 17 (17) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Blood creatinine increased (Investigations) | 5 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood folate decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose abnormal (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose fluctuation (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 17 (17) | 9 (9) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Blood iron decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood magnesium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood potassium increased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure diastolic increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 16 (16) | 8 (8) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Blood pressure systolic increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood sodium increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood testosterone decreased (Investigations) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood thrombin increased (Investigations) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 3 (3)
Blood thyroid stimulating hormone decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood urine present (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Body temperature decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain natriuretic peptide increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 16 (16) | 9 (9) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Sinus arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carbohydrate antigen 19-9 increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac murmur (Investigations) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Chlamydia test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coagulation factor viii level increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coagulation factor increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coagulation test abnormal (Investigations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cortisol decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Creatinine renal clearance increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Crystal urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Culture urine positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ecg signs of ventricular hypertrophy (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram p wave biphasic (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram t wave abnormal (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram t wave amplitude decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram t wave inversion (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Electrocardiogram abnormal (Investigations) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram repolarisation abnormality (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fibrin d dimer increased (Investigations) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 4 (4)
Gamma-glutamyltransferase abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 12 (12) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glucose urine present (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glycosylated haemoglobin increased (Investigations) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiv test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematocrit increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 6 (6) | 9 (9) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio abnormal (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 5 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laboratory test abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipids increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 6 (6) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 9 (9) | 8 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Low density lipoprotein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Mean cell volume decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Monocyte count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mycoplasma test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neisseria test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Norovirus test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oxygen saturation decreased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelet count increased (Investigations) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostatic specific antigen increased (Investigations) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Protein urine present (Investigations) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Prothrombin level increased (Investigations) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Qrs axis abnormal (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Red blood cell count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Red blood cells urine positive (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory rate decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory rate increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Reticulocyte count decreased (Investigations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Reticulocyte count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sars-cov-2 test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serum ferritin decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 11 (11) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Smear cervix abnormal (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Streptococcus test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombin-antithrombin iii complex increased (Investigations) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 2 (2)
Transaminases increased (Investigations) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transferrin saturation increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Troponin i increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Troponin increased (Investigations) | 2 (2) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Urinary casts (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine analysis abnormal (Investigations) | 8 (8) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urine output decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin b1 decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitamin b12 decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitamin d decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 3 (3) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Weight increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cells urine (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cells urine positive (Investigations) | 10 (11) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 3 (3) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Calciphylaxis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 67 (75) | 30 (35) | 14 (14) | 9 (10) | 1 (1) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 11 (11) | 10 (11) | 1 (1) | 1 (1) | 4 (4) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 4 (4) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Folate deficiency (Metabolism and nutrition disorders) | 8 (8) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 8 (8) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 13 (13) | 2 (4) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Histamine intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 18 (18) | 3 (3) | 3 (3) | 5 (6) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 24 (24) | 9 (9) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 6 (6) | 2 (2) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 9 (9) | 9 (9) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Ventricular hypertrophy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 4 (5) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 9 (11) | 3 (3) | 4 (5) | 0 (0) | 2 (2) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (4) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypovitaminosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular hypokinesia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metabolic syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 18 (18) | 8 (8) | 0 (0) | 3 (3) | 2 (2) | 1 (1)
Vitamin b complex deficiency (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vitamin b12 deficiency (Metabolism and nutrition disorders) | 5 (5) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitamin d deficiency (Metabolism and nutrition disorders) | 23 (24) | 10 (10) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Ankle deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 122 (137) | 51 (56) | 16 (19) | 5 (5) | 3 (3) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 9 (9) | 7 (7) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 85 (90) | 53 (57) | 9 (9) | 2 (3) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 7 (8) | 7 (7) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriovenous malformation (Congenital, familial and genetic disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chondromalacia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diastasis recti abdominis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enostosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enthesopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Exostosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femoroacetabular impingement (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermoid cyst (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 11 (11) | 9 (10) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Joint ankylosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint hyperextension (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint noise (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 7 (7) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb mass (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Morphoea (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 22 (22) | 7 (7) | 2 (2) | 1 (1) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-06-13): https://cdn.clinicaltrials.gov/large-docs/25/NCT04625725/Prot_004.pdf
  • Statistical Analysis Plan (2021-07-29): https://cdn.clinicaltrials.gov/large-docs/25/NCT04625725/SAP_005.pdf